CLINICAL TRIAL: NCT02352740
Title: Characterization of the Metabolic Fate of an Oral L-arginine Form in Healthy Subjects Featuring Risk Factors Related to the Metabolic Syndrome.
Brief Title: Characterization of the Metabolic Fate of an Oral Arginine Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Institut de Recherche Pierre Fabre (Other); Hospital Avicenne (Other); Adeprina (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, PU-PH in University Hospitals Paris-Seine-Saint-Denis-APHP-University Hospital Avicenne / Jean Verdier, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: FRMA12-1; 2012-A00755-38 (Other: ANSM)
Record Dates: First submitted 2014-09-24; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Overweight; Hypertriglyceridemic Waist
Keywords: arginine; supplementation; metabolic syndrome; nitric oxide
MeSH Terms: conditions — Overweight; Hypertriglyceridemic Waist; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects with 'hypertriglyceridemic waist' (Experimental): Subjects with overweight, elevated waist circumference and elevated fasting triglyceridemia.
  Intervention : A form arginine and B form arginine
  Interventions: Dietary Supplement: A form Arginine; Dietary Supplement: B form Arginine
- Healthy subjects (Experimental): Control subjects, i.e. without overweight, elevated waist circumference and elevated fasting triglyceridemia.
  Intervention : A form arginine and B form arginine
  Interventions: Dietary Supplement: A form Arginine; Dietary Supplement: B form Arginine

INTERVENTIONS:
Dietary Supplement: A form Arginine — 3 capsules containing 0.5g of A form of L-arginine (1.5g) 3 times daily (4.5g per day) for 1 week
Dietary Supplement: B form Arginine — 3 capsules containing 0.5g of B form of L-arginine (1.5g) 3 times daily (4.5g per day) for 1 week

SUMMARY:
The purpose of this study is to compare the metabolic fate of two oral forms of L-Arginine in healthy subjects featuring metabolic syndrome related risk factors

DETAILED DESCRIPTION:
The study is a randomized crossover study including 16 healthy subjects with risk factors for metabolic syndrome and 16 healthy control subjects. According a double crossover design, each subject received two oral forms of L-arginine (A and B) in random order, and participated in a exploration day on the first day of arginine administration and after one week of supplementation with this arginine form. The two weeks of arginine supplementation were separated by a washout period of 2 weeks at least.

Each exploration extended over 24 hours after administration of the first arginine dose. Blood tests were performed at 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 h after administration of the first dose. During explorations after the supplementation period, we also collected urine (0, 2, 4, 8, 12, 24 h after the first dose).

ELIGIBILITY:
Healthy subjects with 'Hypertriglyceridemic waist' :

Inclusion Criteria:

* Age between 18 to 60 years old
* Overweight (BMI between 25 and 30 kg/m²)
* 'Hypertriglyceridemic waist' (waist circumference > 94cm for men or > 88cm for women and fasting triglyceride levels > 150 mg/dL)

Exclusion Criteria:

* Obesity (BMI> 30 kg / m²)
* Cardiac or vascular diseases
* Diabetes
* Thyroid disease
* Systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg
* Tobacco consumption > 6 cigarettes per week
* Alcohol consumption> 3 drinks per day
* Any medication (except contraceptive treatment) or dietary supplement intake that could not be arrested more than a week before the first visit for the duration of the study.
* Persons under guardianship
* Pregnancy (positive beta-hCG blood test)
* Positive serology HBsAg AcHbc, HCV and HIV
* Hemoglobin < 14 g/dl (for men) or <12 g / dl (for women)
* Participation in a clinical trial within 6 months preceding the study

Healthy control subjects :

Inclusion Criteria:

* Age between 18 to 60 years old
* Normal weight (BMI between 18.5 and 25 kg/m²)
* Waist circumference < 94cm for men or < 88cm for women and fasting triglyceride levels < 150 mg/dL

Exclusion Criteria :

* Cardiac or vascular diseases
* Diabetes
* Thyroid disease
* Systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg
* Tobacco consumption > 6 cigarettes per week
* Alcohol consumption> 3 drinks per day
* Any medication (except contraceptive treatment) or dietary supplement intake that could not be arrested more than a week before the first visit for the duration of the study.
* Persons under guardianship
* Pregnancy (positive beta-hCG blood test)
* Positive serology HBsAg AcHbc, HCV and HIV
* Hemoglobin < 14 g/dl (for men) or <12 g / dl (for women)
* Participation in a clinical trial within 6 months preceding the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Estimate of total conversion of a dose of oral arginine into NO | Repeated measurement for 24h before (day 0) and after supplementation (day 8) for each treatment
  This assessment uses labelled arginine ([15N2-(guanido)]-arginine) for the first dose of arginine taken in the morning, and measurements of 15NO3 in urine for 24h.
  After administration of 15N-arginine, for each urine collection, we determined the nitrate excretion (from measurement of diuresis and nitrate concentration, by reactive chemiluminescence) and isotope 15N enrichment of nitrate ion (by microdiffusion technique and elementary analyzer connected to an isotope mass spectrometerEA-IRMS), to establish, by the principle of isotopic dilution, the total quantities of nitrate specifically from the ingested arginine. The sum of this excretion relative to the ingested dose determined the relative conversion of ingested arginine into NO.
Estimate of kinetic profiles of plasma arginine concentrations over 24 hours | Repeated measurement for 24h before (day 0) and after supplementation (day 8) for each treatment
  Plasma AA concentrations were determined using an ultra-performance liquid chromatography-mass spectrometry system as previously described (Haque and al., 2012).

SECONDARY OUTCOMES:
Quantitative analysis of plasma markers of endothelial function | Before supplementation (day 0) and after supplementation (day 8) for each treatment
  Fasting plasma concentrations of vascular cell adhesion molecule-1 (VCAM-1), intercellular adhesion molecule (ICAM-1), E-Selectin, P-Selectin, Plasminogen activator inhibitor-1 (PAI-1), will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
  In addition, we also have plasma concentrations of nitrite, a marker of of NO production (by reactive chemiluminescence) and other associated markers (3-nitrotyrosine, nitrosothiols, cGMP, in particular ANP, by immunochemistry).
Estimate of kinetics use of arginine for NO and urea synthesis | Repeated measurement for 24h after supplementation (day 8) for each treament
  After administration of 15N-arginine, we measured 15N isotopic enrichment of arginine and citrulline (by mass spectrometry coupled with gas chromatography), of plasma and urinary urea (by separation, by ion exchange, and EA-IRMS) as well as the plasma and urine concentrations in urea. These data and those of arginine and citrulline concentrations provided, by the principle of isotopic dilution, the plasma appearance of ingested arginine and the plasma appearance and urinary excretion of products of its metabolism in NO synthase and arginase ways.
  These data were then subjected to a compartmental modeling work to establish the metabolic flow in these ways.
Other quantitative analysis | Before supplementation (day 0) and after supplementation (day 8) for each treatment
  * Fasting Asymmetric Dimethyl-L-Arginine (ADMA) concentrations were measured by an enzyme-linked immunosorbent assay.
  * The fasting lipid profile (triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol) was measured and were assayed using "classical clinical biochemical analyzers".
  * The fasting insulin and glucose were assayed using "classical clinical biochemical analyzers".
  * Fasting metabolomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, Principal Investigator — Hospital Avicenne; François Mariotti, PhD, Study Director — AgroParisTech
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Background] Abdelhamed AI, Reis SE, Sane DC, Brosnihan KB, Preli RB, Herrington DM. No effect of an L-arginine-enriched medical food (HeartBars) on endothelial function and platelet aggregation in subjects with hypercholesterolemia. Am Heart J. 2003 Mar;145(3):E15. doi: 10.1067/mhj.2003.160. PMID 12660684
- [Background] Adams MR, Forsyth CJ, Jessup W, Robinson J, Celermajer DS. Oral L-arginine inhibits platelet aggregation but does not enhance endothelium-dependent dilation in healthy young men. J Am Coll Cardiol. 1995 Oct;26(4):1054-61. doi: 10.1016/0735-1097(95)00257-9. PMID 7560599
- [Background] Arsenault BJ, Lemieux I, Despres JP, Wareham NJ, Kastelein JJ, Khaw KT, Boekholdt SM. The hypertriglyceridemic-waist phenotype and the risk of coronary artery disease: results from the EPIC-Norfolk prospective population study. CMAJ. 2010 Sep 21;182(13):1427-32. doi: 10.1503/cmaj.091276. Epub 2010 Jul 19. PMID 20643837
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Bai Y, Sun L, Yang T, Sun K, Chen J, Hui R. Increase in fasting vascular endothelial function after short-term oral L-arginine is effective when baseline flow-mediated dilation is low: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2009 Jan;89(1):77-84. doi: 10.3945/ajcn.2008.26544. Epub 2008 Dec 3. PMID 19056561
- [Background] Balkau B, Vernay M, Mhamdi L, Novak M, Arondel D, Vol S, Tichet J, Eschwege E; D.E.S.I.R. Study Group. The incidence and persistence of the NCEP (National Cholesterol Education Program) metabolic syndrome. The French D.E.S.I.R. study. Diabetes Metab. 2003 Nov;29(5):526-32. doi: 10.1016/s1262-3636(07)70067-8. PMID 14631330
- [Background] Beaumier L, Castillo L, Ajami AM, Young VR. Urea cycle intermediate kinetics and nitrate excretion at normal and "therapeutic" intakes of arginine in humans. Am J Physiol. 1995 Nov;269(5 Pt 1):E884-96. doi: 10.1152/ajpendo.1995.269.5.E884. PMID 7491940
- [Background] Berkowitz DE, White R, Li D, Minhas KM, Cernetich A, Kim S, Burke S, Shoukas AA, Nyhan D, Champion HC, Hare JM. Arginase reciprocally regulates nitric oxide synthase activity and contributes to endothelial dysfunction in aging blood vessels. Circulation. 2003 Oct 21;108(16):2000-6. doi: 10.1161/01.CIR.0000092948.04444.C7. Epub 2003 Sep 29. PMID 14517171
- [Background] Blackburn P, Lemieux I, Almeras N, Bergeron J, Cote M, Tremblay A, Lamarche B, Despres JP. The hypertriglyceridemic waist phenotype versus the National Cholesterol Education Program-Adult Treatment Panel III and International Diabetes Federation clinical criteria to identify high-risk men with an altered cardiometabolic risk profile. Metabolism. 2009 Aug;58(8):1123-30. doi: 10.1016/j.metabol.2009.03.012. Epub 2009 Jun 18. PMID 19481769
- [Background] Blackburn P, Lemieux I, Lamarche B, Bergeron J, Perron P, Tremblay G, Gaudet D, Despres JP. Hypertriglyceridemic waist: a simple clinical phenotype associated with coronary artery disease in women. Metabolism. 2012 Jan;61(1):56-64. doi: 10.1016/j.metabol.2011.05.017. Epub 2011 Jul 5. PMID 21733531
- [Background] Blum A, Hathaway L, Mincemoyer R, Schenke WH, Kirby M, Csako G, Waclawiw MA, Panza JA, Cannon RO 3rd. Effects of oral L-arginine on endothelium-dependent vasodilation and markers of inflammation in healthy postmenopausal women. J Am Coll Cardiol. 2000 Feb;35(2):271-6. doi: 10.1016/s0735-1097(99)00553-7. PMID 10676669
- [Background] Bode-Boger SM, Boger RH, Galland A, Tsikas D, Frolich JC. L-arginine-induced vasodilation in healthy humans: pharmacokinetic-pharmacodynamic relationship. Br J Clin Pharmacol. 1998 Nov;46(5):489-97. doi: 10.1046/j.1365-2125.1998.00803.x. PMID 9833603
- [Background] Bode-Boger SM, Muke J, Surdacki A, Brabant G, Boger RH, Frolich JC. Oral L-arginine improves endothelial function in healthy individuals older than 70 years. Vasc Med. 2003 May;8(2):77-81. doi: 10.1191/1358863x03vm474oa. PMID 14518608
- [Background] Bode-Boger SM. Effect of L-arginine supplementation on NO production in man. Eur J Clin Pharmacol. 2006;62:91-9.
- [Background] Boger RH. The pharmacodynamics of L-arginine. J Nutr. 2007 Jun;137(6 Suppl 2):1650S-1655S. doi: 10.1093/jn/137.6.1650S. PMID 17513442
- [Background] Brunner H, Cockcroft JR, Deanfield J, Donald A, Ferrannini E, Halcox J, Kiowski W, Luscher TF, Mancia G, Natali A, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Spieker LE, Taddei S, Webb DJ; Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part II: Association with cardiovascular risk factors and diseases. A statement by the Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Feb;23(2):233-46. doi: 10.1097/00004872-200502000-00001. PMID 15662207
- [Background] Castillo L, Chapman TE, Yu YM, Ajami A, Burke JF, Young VR. Dietary arginine uptake by the splanchnic region in adult humans. Am J Physiol. 1993 Oct;265(4 Pt 1):E532-9. doi: 10.1152/ajpendo.1993.265.4.E532. PMID 8238326
- [Background] Castillo L, deRojas TC, Chapman TE, Vogt J, Burke JF, Tannenbaum SR, Young VR. Splanchnic metabolism of dietary arginine in relation to nitric oxide synthesis in normal adult man. Proc Natl Acad Sci U S A. 1993 Jan 1;90(1):193-7. doi: 10.1073/pnas.90.1.193. PMID 8419922
- [Background] Chan NN, Colhoun HM, Vallance P. Cardiovascular risk factors as determinants of endothelium-dependent and endothelium-independent vascular reactivity in the general population. J Am Coll Cardiol. 2001 Dec;38(7):1814-20. doi: 10.1016/s0735-1097(01)01669-2. PMID 11738279
- [Background] Despres JP, Lemieux I, Bergeron J, Pibarot P, Mathieu P, Larose E, Rodes-Cabau J, Bertrand OF, Poirier P. Abdominal obesity and the metabolic syndrome: contribution to global cardiometabolic risk. Arterioscler Thromb Vasc Biol. 2008 Jun;28(6):1039-49. doi: 10.1161/ATVBAHA.107.159228. Epub 2008 Mar 20. PMID 18356555
- [Background] Fouillet H, Juillet B, Gaudichon C, Mariotti F, Tome D, Bos C. Absorption kinetics are a key factor regulating postprandial protein metabolism in response to qualitative and quantitative variations in protein intake. Am J Physiol Regul Integr Comp Physiol. 2009 Dec;297(6):R1691-705. doi: 10.1152/ajpregu.00281.2009. Epub 2009 Oct 7. PMID 19812354
- [Background] Gomez-Huelgas R, Bernal-Lopez MR, Villalobos A, Mancera-Romero J, Baca-Osorio AJ, Jansen S, Guijarro R, Salgado F, Tinahones FJ, Serrano-Rios M. Hypertriglyceridemic waist: an alternative to the metabolic syndrome? Results of the IMAP Study (multidisciplinary intervention in primary care). Int J Obes (Lond). 2011 Feb;35(2):292-9. doi: 10.1038/ijo.2010.127. Epub 2010 Jun 15. PMID 20548300
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; National Heart, Lung, and Blood Institute; American Heart Association. Definition of metabolic syndrome: report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Arterioscler Thromb Vasc Biol. 2004 Feb;24(2):e13-8. doi: 10.1161/01.ATV.0000111245.75752.C6. No abstract available. PMID 14766739
- [Background] Hill BG, Dranka BP, Bailey SM, Lancaster JR Jr, Darley-Usmar VM. What part of NO don't you understand? Some answers to the cardinal questions in nitric oxide biology. J Biol Chem. 2010 Jun 25;285(26):19699-704. doi: 10.1074/jbc.R110.101618. Epub 2010 Apr 21. PMID 20410298
- [Background] Joshi MS, Ferguson TB Jr, Johnson FK, Johnson RA, Parthasarathy S, Lancaster JR Jr. Receptor-mediated activation of nitric oxide synthesis by arginine in endothelial cells. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):9982-7. doi: 10.1073/pnas.0506824104. Epub 2007 May 29. PMID 17535904
- [Background] Kim JA, Montagnani M, Koh KK, Quon MJ. Reciprocal relationships between insulin resistance and endothelial dysfunction: molecular and pathophysiological mechanisms. Circulation. 2006 Apr 18;113(15):1888-904. doi: 10.1161/CIRCULATIONAHA.105.563213. PMID 16618833
- [Background] Lauer T, Heiss C, Balzer J, Kehmeier E, Mangold S, Leyendecker T, Rottler J, Meyer C, Merx MW, Kelm M, Rassaf T. Age-dependent endothelial dysfunction is associated with failure to increase plasma nitrite in response to exercise. Basic Res Cardiol. 2008 May;103(3):291-7. doi: 10.1007/s00395-008-0714-3. Epub 2008 Mar 17. PMID 18347836
- [Background] Lee J, Ryu H, Ferrante RJ, Morris SM Jr, Ratan RR. Translational control of inducible nitric oxide synthase expression by arginine can explain the arginine paradox. Proc Natl Acad Sci U S A. 2003 Apr 15;100(8):4843-8. doi: 10.1073/pnas.0735876100. Epub 2003 Mar 24. PMID 12655043
- [Background] Li H, Forstermann U. Prevention of atherosclerosis by interference with the vascular nitric oxide system. Curr Pharm Des. 2009;15(27):3133-45. doi: 10.2174/138161209789058002. PMID 19754387
- [Background] Loscalzo J. What we know and don't know about L-arginine and NO. Circulation. 2000 May 9;101(18):2126-9. doi: 10.1161/01.cir.101.18.2126. No abstract available. PMID 10801749
- [Background] Luiking YC, Engelen MP, Deutz NE. Regulation of nitric oxide production in health and disease. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):97-104. doi: 10.1097/MCO.0b013e328332f99d. PMID 19841582
- [Background] Maas R, Schwedhelm E, Kahl L, Li H, Benndorf R, Luneburg N, Forstermann U, Boger RH. Simultaneous assessment of endothelial function, nitric oxide synthase activity, nitric oxide-mediated signaling, and oxidative stress in individuals with and without hypercholesterolemia. Clin Chem. 2008 Feb;54(2):292-300. doi: 10.1373/clinchem.2007.093575. Epub 2007 Dec 10. PMID 18070819
- [Background] Mariotti F, Mahe S, Luengo C, Benamouzig R, Tome D. Postprandial modulation of dietary and whole-body nitrogen utilization by carbohydrates in humans. Am J Clin Nutr. 2000 Oct;72(4):954-62. doi: 10.1093/ajcn/72.4.954. PMID 11010937
- [Background] Mariotti F, Huneau JF, Szezepanski I, Petzke KJ, Aggoun Y, Tome D, Bonnet D. Meal amino acids with varied levels of arginine do not affect postprandial vascular endothelial function in healthy young men. J Nutr. 2007 Jun;137(6):1383-9. doi: 10.1093/jn/137.6.1383. PMID 17513395
- [Background] Mariotti F, Petzke KJ, Bonnet D, Szezepanski I, Bos C, Huneau JF, Fouillet H. Kinetics of the utilization of dietary arginine for nitric oxide and urea synthesis: insight into the arginine-nitric oxide metabolic system in humans. Am J Clin Nutr. 2013 May;97(5):972-9. doi: 10.3945/ajcn.112.048025. Epub 2013 Mar 27. PMID 23535108
- [Background] Mariotti F, Huneau JF, Petzke KJ, Szezepanski I, Tomé D, Bos C, Bonnet D. Malgré une assez forte extraction splanchnique pour l'uréogenèse, l'arginine alimentaire, à dose nutritionnelle, est largement, et de façon dose-dépendante, disponible pour les tissus périphériques. Nutr Clin Metab. 2008:22(S1):5.
- [Background] Maxwell AJ. Mechanisms of dysfunction of the nitric oxide pathway in vascular diseases. Nitric Oxide. 2002 Mar;6(2):101-24. doi: 10.1006/niox.2001.0394. PMID 11890735
- [Background] Moncada S, Higgs EA. Molecular mechanisms and therapeutic strategies related to nitric oxide. FASEB J. 1995 Oct;9(13):1319-30. PMID 7557022
- [Background] Moncada S, Higgs EA. The discovery of nitric oxide and its role in vascular biology. Br J Pharmacol. 2006 Jan;147 Suppl 1(Suppl 1):S193-201. doi: 10.1038/sj.bjp.0706458. PMID 16402104
- [Background] Morris SM Jr. Recent advances in arginine metabolism: roles and regulation of the arginases. Br J Pharmacol. 2009 Jul;157(6):922-30. doi: 10.1111/j.1476-5381.2009.00278.x. Epub 2009 Jun 5. PMID 19508396
- [Background] Napoli C, de Nigris F, Williams-Ignarro S, Pignalosa O, Sica V, Ignarro LJ. Nitric oxide and atherosclerosis: an update. Nitric Oxide. 2006 Dec;15(4):265-79. doi: 10.1016/j.niox.2006.03.011. Epub 2006 Apr 15. PMID 16684613
- [Background] Nawabzad R, Champin B. [Concordance between three definitions for metabolic syndrome (Hypertriglyceridemic waist, National Cholesterol Education Program, International Diabetes Federation), and prevalence of the syndrome in a French population]. Rev Prat. 2010 Dec 20;60(10 Suppl):15-23. French. PMID 22530271
- [Background] Ohta F, Takagi T, Sato H, Ignarro LJ. Low-dose L-arginine administration increases microperfusion of hindlimb muscle without affecting blood pressure in rats. Proc Natl Acad Sci U S A. 2007 Jan 23;104(4):1407-11. doi: 10.1073/pnas.0610207104. Epub 2007 Jan 17. PMID 17229841
- [Background] Preli RB, Klein KP, Herrington DM. Vascular effects of dietary L-arginine supplementation. Atherosclerosis. 2002 May;162(1):1-15. doi: 10.1016/s0021-9150(01)00717-1. PMID 11947892
- [Background] Rizzo NO, Maloney E, Pham M, Luttrell I, Wessells H, Tateya S, Daum G, Handa P, Schwartz MW, Kim F. Reduced NO-cGMP signaling contributes to vascular inflammation and insulin resistance induced by high-fat feeding. Arterioscler Thromb Vasc Biol. 2010 Apr;30(4):758-65. doi: 10.1161/ATVBAHA.109.199893. Epub 2010 Jan 21. PMID 20093624
- [Background] Schafer A, Wiesmann F, Neubauer S, Eigenthaler M, Bauersachs J, Channon KM. Rapid regulation of platelet activation in vivo by nitric oxide. Circulation. 2004 Apr 20;109(15):1819-22. doi: 10.1161/01.CIR.0000126837.88743.DD. Epub 2004 Apr 5. PMID 15066953
- [Background] Schwedhelm E, Maas R, Freese R, Jung D, Lukacs Z, Jambrecina A, Spickler W, Schulze F, Boger RH. Pharmacokinetic and pharmacodynamic properties of oral L-citrulline and L-arginine: impact on nitric oxide metabolism. Br J Clin Pharmacol. 2008 Jan;65(1):51-9. doi: 10.1111/j.1365-2125.2007.02990.x. Epub 2007 Jul 27. PMID 17662090
- [Background] Siani A, Pagano E, Iacone R, Iacoviello L, Scopacasa F, Strazzullo P. Blood pressure and metabolic changes during dietary L-arginine supplementation in humans. Am J Hypertens. 2000 May;13(5 Pt 1):547-51. doi: 10.1016/s0895-7061(99)00233-2. PMID 10826408
- [Background] Siekmeier R, Grammer T, Marz W. Roles of oxidants, nitric oxide, and asymmetric dimethylarginine in endothelial function. J Cardiovasc Pharmacol Ther. 2008 Dec;13(4):279-97. doi: 10.1177/1074248408326488. Epub 2008 Oct 22. PMID 18945874
- [Background] Siervo M, Jackson SJ, Bluck LJ. In-vivo nitric oxide synthesis is reduced in obese patients with metabolic syndrome: application of a novel stable isotopic method. J Hypertens. 2011 Aug;29(8):1515-27. doi: 10.1097/HJH.0b013e3283487806. PMID 21720276
- [Background] Siervo M, Stephan BC, Feelisch M, Bluck LJ. Measurement of in vivo nitric oxide synthesis in humans using stable isotopic methods: a systematic review. Free Radic Biol Med. 2011 Aug 15;51(4):795-804. doi: 10.1016/j.freeradbiomed.2011.05.032. Epub 2011 Jun 13. PMID 21672626
- [Background] Tangphao O, Grossmann M, Chalon S, Hoffman BB, Blaschke TF. Pharmacokinetics of intravenous and oral L-arginine in normal volunteers. Br J Clin Pharmacol. 1999 Mar;47(3):261-6. doi: 10.1046/j.1365-2125.1999.00883.x. PMID 10215749
- [Background] Tousoulis D, Kampoli AM, Tentolouris C, Papageorgiou N, Stefanadis C. The role of nitric oxide on endothelial function. Curr Vasc Pharmacol. 2012 Jan;10(1):4-18. doi: 10.2174/157016112798829760. PMID 22112350
- [Background] Tsikas D, Boger RH, Sandmann J, Bode-Boger SM, Frolich JC. Endogenous nitric oxide synthase inhibitors are responsible for the L-arginine paradox. FEBS Lett. 2000 Jul 28;478(1-2):1-3. doi: 10.1016/s0014-5793(00)01686-0. PMID 10922458
- [Background] Voetsch B, Jin RC, Loscalzo J. Nitric oxide insufficiency and atherothrombosis. Histochem Cell Biol. 2004 Oct;122(4):353-67. doi: 10.1007/s00418-004-0675-z. Epub 2004 Aug 26. PMID 15338226
- [Background] West SG, Likos-Krick A, Brown P, Mariotti F. Oral L-arginine improves hemodynamic responses to stress and reduces plasma homocysteine in hypercholesterolemic men. J Nutr. 2005 Feb;135(2):212-7. doi: 10.1093/jn/135.2.212. PMID 15671215
- [Background] Wilkinson IB, Qasem A, McEniery CM, Webb DJ, Avolio AP, Cockcroft JR. Nitric oxide regulates local arterial distensibility in vivo. Circulation. 2002 Jan 15;105(2):213-7. doi: 10.1161/hc0202.101970. PMID 11790703
- [Background] Wu G, Morris SM Jr. Arginine metabolism: nitric oxide and beyond. Biochem J. 1998 Nov 15;336 ( Pt 1)(Pt 1):1-17. doi: 10.1042/bj3360001. PMID 9806879
- [Background] Wu G, Meininger CJ. Arginine nutrition and cardiovascular function. J Nutr. 2000 Nov;130(11):2626-9. doi: 10.1093/jn/130.11.2626. PMID 11053497
- [Background] Wu G, Meininger CJ. Regulation of nitric oxide synthesis by dietary factors. Annu Rev Nutr. 2002;22:61-86. doi: 10.1146/annurev.nutr.22.110901.145329. Epub 2002 Jan 4. PMID 12055338
- [Background] Wyatt AW, Steinert JR, Mann GE. Modulation of the L-arginine/nitric oxide signalling pathway in vascular endothelial cells. Biochem Soc Symp. 2004;(71):143-56. doi: 10.1042/bss0710143. PMID 15777019
- [Background] Yang Z, Ming XF. Recent advances in understanding endothelial dysfunction in atherosclerosis. Clin Med Res. 2006 Mar;4(1):53-65. doi: 10.3121/cmr.4.1.53. PMID 16595793
- [Derived] Deveaux A, Fouillet H, Petzke KJ, Hermier D, Andre E, Bunouf P, Lantoine-Adam F, Benamouzig R, Mathe V, Huneau JF, Mariotti F. A Slow- Compared with a Fast-Release Form of Oral Arginine Increases Its Utilization for Nitric Oxide Synthesis in Overweight Adults with Cardiometabolic Risk Factors in a Randomized Controlled Study. J Nutr. 2016 Jul;146(7):1322-9. doi: 10.3945/jn.116.231910. Epub 2016 Jun 8. PMID 27281799